CLINICAL TRIAL: NCT06330844
Title: Race Based Stress and Empowerment Focused Compensatory Cognitive Training for Mild Cognitive Impairment
Brief Title: Race-Based Stress and Cognitive Training for MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Rachael Ellison, Principle Investigator, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBSEF-MCI-CCT
Record Dates: First submitted 2024-02-09; First posted 2024-03-26 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two groups assignment - One group will complete the original ME-CCT training program. The other group will complete the newly developed RBSE-CCT-MCI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: RBSEF-CCT-MCI (Experimental): Participants will complete the newly developed RBSE-CCT-MCI training program.
  Interventions: Behavioral: Race Based Stress and Empowerment Focused Compensatory Cognitive Training for Mild Cognitive Impairment (RBSEF-CCT-MCI)
- Control Group: ME-CCT (Other): Participants will complete the original, ME-CCT training program.
  Interventions: Behavioral: Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment (ME-CCT)

INTERVENTIONS:
Behavioral: Race Based Stress and Empowerment Focused Compensatory Cognitive Training for Mild Cognitive Impairment (RBSEF-CCT-MCI) — RBSEF-CCT-MCI differs from ME-CCT in that this intervention integrates psychoeducation and strategies for processing and coping with race/ethnicity-related stressors, as part of the larger conversation in ME-CCT regarding stress, and how stress interferes with attention, learning, and subsequently one's subjective sense of memory.
  Arms: Experimental: RBSEF-CCT-MCI
Behavioral: Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment (ME-CCT) — ME-CCT focuses on:
  1. Cognitive training, psychotherapeutic, and lifestyle techniques.
  2. Incorporates CCT techniques designed to help patients manage problems with memory, attention, and executive functions (i.e., organization, planning, decision-making, and problem-solving).
  3. Includes mindfulness-based stress reduction practice which has been shown to improve cognitive and neuropsychiatric function in various populations.
  Arms: Control Group: ME-CCT

SUMMARY:
This a two phase project that aims to pilot a new adaptation (Phase 1) of Motivationally Enhanced Compensatory Cognitive Training for Mild Cognitive Impairment (ME-CCT; an originally VA-based cognitive rehabilitation manualized intervention for older adults with MCI, with a focus on the impact of stress on cognitive functioning; that integrates components from the Race Based Stress and Empowerment (RBSE) group for an increased focus on race-based stress and discrimination for racial minority older adults (i.e., RBSEF-CCT-MCI). In a pilot open trial, 75-150 participants will receive group-based intervention for 8 weeks, with 8-10 participants per group.

Following the pilot study, the investigators will complete a randomized controlled trial (RCT) (Phase 2) to compare the efficacy of the RBSEF-CCT-MCI with the ME-CCT. In the RCT, 75-150 participants will be randomized into either 1) The active control group, who will complete the original, ME-CCT training program, or 2) The experimental group, who will complete the newly developed RBSE-CCT-MCI. Both research groups will complete the interventions for 8 weeks, with 8-10 participants per group.

Hypothesis: Participation in this newly developed/updated intervention (i.e., RBSEF-CCT-MCI) will result in improvements in both (a) subjective and (b) objective cognitive functioning, and (c) self-reported mental health symptoms.

DETAILED DESCRIPTION:
African American (AA) individuals are at higher risk for non-normative cognitive decline, particularly due to increased rates of cardiovascular and cerebrovascular risk factors. These types of risk factors (e.g., hypertension, diabetes mellitus, obesity, hyperlipidemia, etc.) are independently associated with brain imaging changes, even before potential clinical manifestation of cardiovascular or cerebrovascular disease.

When compared to the general aging population, AA adults experience disproportionately higher rates of hypertension as well as both an earlier age of onset and higher concomitant morbidity and mortality from hypertension when compared to any other racial/ethnic group in the US. AA individuals experience greater exposure to specific chronic stressors, such as discrimination and low socioeconomic status, as well as report higher overall levels of stress compared to white individuals. However, racial disparities in hypertension rates persist even after controlling for socioeconomic status. Researchers have failed to demonstrate any risk factors that are biologically unique to AA patients. These findings have led researchers to consider other psychosocial and environmental factors that may explain the observed hypertension disparities, namely, racial discrimination and racial segregation.

AA older adults are not only at higher risk for non-normative cognitive decline due to both semi-direct (i.e., increased risk of cardiovascular/cerebrovascular risk factors, such as HTN), but other factors such as race-related stress may not only exacerbate these risk factors, but also interfere day-to-day with optimal cognitive performance due to overall increased stress and diversion of cognitive resources. Therefore, for AA older adults, there is an increased need not only for interventions that help to compensate for cognitive decline and increase daily functioning, but also an increased need for an intervention to reduce the effects of race-related stressors. The proposed Race-Based Stress and Empowerment Focused Compensatory Cognitive Training for Mild Cognitive Impairment (RBSEF-CCT-MCI) as proposed in this pilot, is one such intervention that would accomplish those aims and has the potential for a significant impact on patient care for AA older adults who could benefit from additional tools and strategies to improve cognitive functioning and increase day-to-day independent functioning.

Of note, original authors of both protocols have granted consent for modifications of their interventions, and the investigators already have a draft of the new protocol.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted in-person, so they must be able to travel to Rosalind Franklin University.
* The study will initially be limited to participants who self-identify as Black/African American, or who self-identify with other racial/ethnic groups in addition to self-identifying as Black/African-American; however, may be expanded to include participants that identify as Hispanic/Latine.

Exclusion Criteria:

* Participants are ineligible to participate in this study if they are not at least 65 years of age and are not experiencing at least mild cognitive impairment or self-reported cognitive difficulties.
* Participants will also be excluded if they have a diagnosis of dementia (i.e., major neurocognitive disorder), intellectual disability, mild head injury (i.e., concussion) within the last six months, and/or a history of moderate to severe traumatic brain injury.
* Diagnosis of dementia may be from self-report or other medical records, or for participants to fail screening cognitive assessments (i.e., the RBANS) that would suggest they may be at the level of dementia (i.e., major neurocognitive disorder) as ultimately determined by study PI with objective scores less then 2 standard deviations below the mean on the RBANS.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Verbal learning and memory | up to eight weeks
  Assessed by the California Verbal Learning Test- Second Edition (CVLT-II)
Basic auditory attention and working memory | up to eight weeks
  Assessed by the Digit Span subtest of the Wechsler Adult Intelligence Scale (WAIS-IV)
Psychomotor processing speed | up to eight weeks
  Assessed by the Coding and Symbol search subtests of the WAIS-IV
Psychomotor processing speed; executive functioning | up to eight weeks
  As assessed by the Stroop Test
Self-report of prospective and retrospective memory | up to eight weeks
  The Prospective and Retrospective Memory Questionnaire (PRMQ). The PRMQ developed to provide a self-report measure of prospective and retrospective memory slips in everyday life. It consists of sixteen items, eight asking about prospective memory failures, and eight concerning retrospective failures.
Self-report of cognitive concerns | up to eight weeks
  Neuro-QOL (neuro-quality of life); applied cognition: general concerns & executive functioning (EF) subscales
The Patient Health Questionnaire-9 | up to eight weeks
  (i.e., PHQ-9; assessing self-report symptoms of depression)
Self-report symptoms of anxiety | up to eight weeks
  As assessed by the Generalized Anxiety Disorder-7 questionnaire (i.e., GAD-7)
Self-reported daily functioning | up to eight weeks
  As assessed by The World Health Organization Disability Assessment Schedule 2.0 (i.e., WHODAS 2.0)
The Racial Microaggressions Scale | up to eight weeks
  Assessing the occurrence and distress elicited by racial indignities, slights, mistreatment, or offenses that people of color may face on a recurrent or consistent basis.
The Trauma Symptoms of Discrimination Scale | up to eight weeks
  Self-report measure assessing the traumatizing impact of discrimination broadly by measuring anxiety-related symptoms of trauma due to discriminatory experiences

CONTACTS AND LOCATIONS:
Overall Officials: Rachael L Ellison, PhD, Principal Investigator — Rosalind Franklin University of Medicine and Science
Locations (1):
- Rosalind Franklin University of Medicine and Science, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huckans M, Hutson L, Twamley E, Jak A, Kaye J, Storzbach D. Efficacy of cognitive rehabilitation therapies for mild cognitive impairment (MCI) in older adults: working toward a theoretical model and evidence-based interventions. Neuropsychol Rev. 2013 Mar;23(1):63-80. doi: 10.1007/s11065-013-9230-9. Epub 2013 Mar 8. PMID 23471631
- [Background] Nayak US. Design participation by the thousand elders. Stud Health Technol Inform. 1998;48:423-7. No abstract available. PMID 10186562
- [Background] Kremer A, Focaccia G, Ferreyra R, Kraly A, Sniechowski T. [The epidemiology of cancer in the Province of Neuquen, Argentina]. Medicina (B Aires). 1987;47(5):471-6. No abstract available. Spanish. PMID 3504986
- [Background] Fritsch J, Wolf P. [Cog-rail extension corset in the surgical management of scoliosis]. Beitr Orthop Traumatol. 1973 Feb;20(2):124-7. No abstract available. German. PMID 4700211
- [Background] Spruill TM, Butler MJ, Thomas SJ, Tajeu GS, Kalinowski J, Castaneda SF, Langford AT, Abdalla M, Blackshear C, Allison M, Ogedegbe G, Sims M, Shimbo D. Association Between High Perceived Stress Over Time and Incident Hypertension in Black Adults: Findings From the Jackson Heart Study. J Am Heart Assoc. 2019 Nov 5;8(21):e012139. doi: 10.1161/JAHA.119.012139. Epub 2019 Oct 16. PMID 31615321
- [Background] Inoue S. Uptake of 3-H-DL-leucine and 3-H-uridine by the caudal neurosecretory system of the loach (Misgurnus anguillicaudatus) maintained in vitro. Endocrinol Jpn. 1968 Dec;15(4):505-7. doi: 10.1507/endocrj1954.15.505. No abstract available. PMID 5756074